CLINICAL TRIAL: NCT06541444
Title: An Open, Single Center Exploratory Study to Evaluate Safety and Efficacy of NK520 for Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Safety and Efficacy of NK520 to Treat Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Base Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NK520-02
Record Dates: First submitted 2024-06-07; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A(low-dose group) (Experimental): NK520: 3×10^7NK/kg
  Interventions: Drug: NK520
- Group B(medium-dose group) (Experimental): NK520: 6×10^7NK/kg
  Interventions: Drug: NK520
- Group C(high-dose group) (Experimental): NK520: 9×10^7NK/kg
  Interventions: Drug: NK520

INTERVENTIONS:
Drug: NK520 — The number of NK520 cell infused for each dosing will be calculated based on body weight of subject. NK520 should be administered through intravenous infusion once a week, for a total of four times.
  Other Names: genetic modified NK cell

SUMMARY:
This study will evaluate the safety and efficacy of NK520 in the treatment of relapsed/refractory acute myeloid leukemia. NK520 will be administered by intravenous injection. The safety and efficacy of this treatment will be evaluated.

DETAILED DESCRIPTION:
This open label, single-arm study aims to evaluate the efficacy and safety of allogenic NK cells in subjects with relapsed/refractory acute myeloid leukemia. Allogenic NK cells will be infused once a week. After infusion, the investigators will observe the characteristics of dose limited toxicity (DLT), and determine the maximum tolerable dose(MTD). To provide basis for the dosage and treatment plan of cell products in follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between 18 and 75 years;
2. Diagnostic Criteria:

   Meet the 2016 World Health Organization (WHO) diagnostic criteria for AML, unsuitable for current treatments or patients with relapsed/refractory AML after ≥2 lines of therapy. The definition of relapsed/refractory acute myeloid leukemia is based on the 2017 Chinese Guidelines for Diagnosis and Treatment:
   1. Relapsed AML: Diagnosis is confirmed when leukemia cells reappear in the peripheral blood or bone marrow blast cells exceed 5% after complete remission (CR) (excluding reasons such as bone marrow regeneration post-consolidation chemotherapy) or there is extramedullary infiltration by leukemia cells;
   2. Refractory AML: Initial cases unresponsive after two cycles of standard regimen treatment; recurrence within 12 months after CR and consolidation therapy; recurrence beyond 12 months with ineffectiveness of conventional chemotherapy; those who have relapsed twice or more; or persistent extramedullary leukemia;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
4. Expected survival of at least 12 weeks;
5. Normal Organ Function.

Exclusion Criteria:

1. Acute promyelocytic leukemia;
2. Severe bleeding tendency or coagulation disorders, or currently receiving thrombolytic therapy;
3. Active tuberculosis (TB), currently undergoing anti-TB treatment, or treated for TB within 1 year prior to the study;
4. HIV-infected individuals, or known active syphilis infection;
5. Use of immunosuppressive drugs within 1 week before the first dose, excluding topical, inhaled, or other locally administered glucocorticoids, or physiologic doses of systemic glucocorticoids (not exceeding 10 mg/day prednisone equivalent) for allergic reactions or for managing respiratory distress from asthma, COPD, etc;
6. Receipt of live attenuated vaccines within 2 weeks before the first dose or planned during the study;
7. Participation in another clinical trial and receipt of investigational drug within 4 weeks prior to the first dose;
8. Receipt of immune-modulating drugs (including thymosin, interferons, except for local use to control pleural or ascitic fluid) within 2 weeks prior to the first dose;
9. At screening, hepatitis B or C viral tests positive according to either:

   * HBsAg positive with serum HBV-DNA titer ≥1×10^3 copies/mL or above normal limits;
   * HCV antibody positive;
10. Any other condition or situation in which the investigator deems the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | From the first dose of NK520 to 4 weeks after last infusion of NK520
  To evaluate the DLT during NK520 treatment
Complete Response Rate (CRR) | From the date of first infusion of NK520 up to 104 weeks.
  Effectiveness Metrics

SECONDARY OUTCOMES:
Overall response rate (ORR) | From the date of first infusion of NK520 up to 104 weeks.
  Effectiveness Metrics
Event-Free Survival (EFS) | From date of enrollment up to 104 weeks, or date of progression, or date of death, whichever came first.
  Effectiveness Metrics
Overall Survival (OS) | From date of enrollment up to 104 weeks or date of death, whichever came first.
  Effectiveness Metrics
Duration of Response (DOR) | From the date of enrollment up to 104 weeks
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Overall Officials: zhiguo Long, Principal Investigator — Shanghai Pudong Hospital
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No